CLINICAL TRIAL: NCT04517409
Title: Goal-directed Hemodynamic Therapy Based on Stroke Volume, Pulse Pressure Variation and Continuosus Cardiac Index in Patiens Undergoing Major Hepatic Resection
Brief Title: Goal-directed Hemodynamic Therapy in Patiens Undergoing Major Hepatic Resection
Acronym: GOAL-HEMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Castilla-La Mancha Health Service (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 4161
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Hemodynamic Monitoring

STUDY DESIGN:
Intervention Model Description: Prospective randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GDHT (Experimental): After hepatic resection (Dynamic phase), the patients received an initial hemodynamic assessment based on PPV, CI and MAP. First, preload was optimized by fluid loading until PPV was <14% or VVS <12%, subjects were given 4 ml kg-1 boluses colloid solution every 5 minutes. At this point, the patient's individual preload optimized CI was determined and used as the hemodynamic goal until the end of surgery. Only if this value was below 2.5 L/min/(m2), inotropes were applied to reach this minimum CI, serving as a safety parameter to prevent patients from low cardiac output. If PPV and CI were within the target range but MAP was below 65 mmHg or PPV/VVS>1,2, vasopressors were started. After the initial assessment, patients were reassessed every 15 minutes intraoperatively to maintain values.
  Interventions: Procedure: Goal-directed hemodynamic therapy
- Control (Other): Before hepatic resection (Static phase) all patiens received continuous infusion of balanced crystalloid with the goal of CVP of 5 mmHg.
  After hepatic resection (Dynamic phase), the patiens received colloid solution, vasopressors, and inotropes at the discretion of the anaesthetist, acording to CVP, MAP and orine output. In this group, CO monitoring was not performed. Intraoperative treatment goals in the control arm were flexible to avoid both extremes of clinical practice and practice misalignment
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Goal-directed hemodynamic therapy — Eligible patients were equally randomized into two study groups: 1) Standard perioperative (Control group ) and 2) hemodinamic management based using radial artery pulse contour analysis (GDHT group). Randomization was performed the day before surgery by the study member responsable for anesthesia delivery using sealed opaque envelope technique stored in non-transparent containers with group allocation in a 1:1 ratio. Only patients were blinded to group allocation. Care providers and investigators could not be blinded due to the presence of the cardiac index trending monitor
  Other Names: GDHT
  Arms: GDHT
Procedure: Control — Before hepatic resection (Static phase) all patiens received continuous infusion of balanced crystalloid with the goal of CVP of 5 mmHg.
  After hepatic resection (Dynamic phase), the patiens received colloid solution, vasopressors, and inotropes at the discretion of the anaesthetist, acording to CVP, MAP and orine output. In this group, CO monitoring was not performed. Intraoperative treatment goals in the control arm were flexible to avoid both extremes of clinical practice and practice misalignment.
  Arms: Control

SUMMARY:
The aim of the study of patients undergoing major hepatic resection was compared standard perioperative (control Group) with hemodinamic management based on PPV, VVS, continuos CO trending and dynamic arterial elastance using radial artery pulse contour analysis (GDHT group). We hypothessized that following this treatment regimen after hepatic resection results in reduced postoperative complications (primary endpoint) and reduced length of hospital stay (secundary endpoint)

DETAILED DESCRIPTION:
The study was performed as a prospective randomized trial at the Department of Anesthesiology and Intensive Care Medicine and the Department of Surgery of the Hospital Universitario de Ciudad Real, Spain.Faculty. The study was approved by the local ethical committee. All patients scheduled for hepatic resection of more than two segments were found eligible for study inclusion. Exclusion criteria were: age less than 18, body weight less than 50 kg or more than 150 kg, irregular heart rhythm, severe cardiovascular disease (chronic heart failure, valvular abnormality, cardiomyopathy, etc.), severe liver dysfunction (Child Pugh score B or C). All participants signed informed consent prior study inclusion.

Protocol of the study.

Eligible patients were equally randomized into two study groups: 1) Standard perioperative (Control group ) and 2) hemodinamic management based using radial artery pulse contour analysis (GDHT group). Randomization was performed the day before surgery by the study member responsable for anesthesia delivery using sealed opaque envelope technique stored in non-transparent containers with group allocation in a 1:1 ratio. Only patients were blinded to group allocation. Care providers and investigators could not be blinded due to the presence of the cardiac index trending monitor.

Intraoperative management.

All subjects received balanced anaesthesia, i.v. anaesthetic induction, and neuromuscular relaxants; for pragmatic reasons, their administration was at the discretion of the anaesthetist. Bispectral index monitoring was used to monitor the depth of anaesthesia. Sevoflurane was used for anaesthesia maintenance, with a BIS target range of 40-60. Central venous catheter placement and invasive radial arterial blood pressure monitoring were performed per preference of the anaesthetist.

All subjects had basic anaesthetic monitoring with fivelead ECG, pulse oximetry, and oscillometric blood pressure; at least one peripheral i.v. line was established. All subjects received standard measures to maintain oxygen saturation by pulse oximetry >94%, normothermia, and heart rate <100 beats min-1. Ventilation with inspired oxygen fraction of 60% was mechanically controlled to maintain PaCO2 between 4.7 and 6.0 kPa, with a positive end-expiratory pressure of 4-6mm Hg and tidal volume of 6-8 ml kg-1.

In cases when PM was used, hemodynamic data were recorded one minute before the clamp, one minute after the clamp and one minute afterthe PM's release. Ephedrine was given in case of hemodynamic instability (mean arterial pressure <65 mmHg) and if repeated boluses were ineffective, noradrenaline infusion was started.

In a case of acute blood loss (more than 150 mL/ min or more than 500 mL), colloid infusion of was administered with respect to maximal recommended dose (30 mL/kg).

In both groups, blood loss was compensated for by infusión of colloid in a 1:1 ratio. Packed red cells were transfused for haemoglobin <10 g dl-1 in subjects with cardiac comorbidities, or <7 g dl-1 in those without cardiac comorbidities.

Hemodynamic data were documented every 15 minutes. At the beginning of hepatic resection, middle and at the end of surgery blood samples were drawn for arterial and central venous blood gas analysis. At the end of surgery total catecholamine administration, estimated blood loss, urine output and infused fluids were recorded. The time between the end of surgery and extubation was recorded.

GDHT group.

The arterial line was additionally connected to the cardiac index trending monitor (ProAQT, PULSION Medical Systems SE, Munich, Germany).

Fluid therapy was given. Before hepatic resection (Static phase) all patiens received continuous infusion of balanced crystalloid fluids (Ringer,s lactate) at 1 ml kg-1h-1 After hepatic resection (Dynamic phase), the patients received an initial hemodynamic assessment based on PPV, CI and MAP, as shown in Figure 1. First, preload was optimized by fluid loading until PPV was <14% or VVS <12%, subjects were given 4 ml kg-1 boluses colloid solution every 5 minutes. At this point, the patient's individual preload optimized CI was determined and used as the hemodynamic goal until the end of surgery. Only if this value was below 2.5 L/min/(m2), inotropes were applied to reach this minimum CI, serving as a safety parameter to prevent patients from low cardiac output. If PPV and CI were within the target range but MAP was below 65 mmHg or PPV/VVS>1,2, vasopressors were started. After the initial assessment, patients were reassessed every 15 minutes intraoperatively to maintain values

ELIGIBILITY:
Inclusion Criteria:

All patients scheduled for hepatic resection of more than two segments

Exclusion Criteria:

age less than 18, body weight less than 50 kg or more than 150 kg, irregular heart rhythm, severe cardiovascular disease (chronic heart failure, valvular abnormality, cardiomyopathy, etc.), severe liver dysfunction (Child Pugh score B or C).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-11-05 (Actual); Primary Completion 2017-11-05 (Actual); Study Completion 2017-11-05 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 180 days
  Pre-defined postoperative complications for each patient were recorded after surgery from the patient record and by visiting patients on the ward by the investigators

IPD SHARING:
Plan to Share IPD: Undecided